CLINICAL TRIAL: NCT00685165
Title: A Randomized, Two-Way, Single-Dose, Open-Label Study to Evaluate the Bioequivalence of a Test Tablet Formulation of Primidone 50 mg, Compared to an Equivalent Dose of Primidone (Mysoline®) in Healthy Adult Subjects
Brief Title: Fasted Bioequivalence Study of Primidone Tablets and Mysoline Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Kristin Arnold, Vice President R&D, Mutual Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 04090
Record Dates: First submitted 2008-05-24; First posted 2008-05-28 (Estimated); Results first posted 2010-01-20 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-11

CONDITIONS: Therapeutic Equivalency
MeSH Terms: interventions — Primidone; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primidone 50 mg Tablets (Experimental): A single dose of primidone 50 mg administered after an overnight fast of at least 10 hours.
  Interventions: Drug: Primidone 50 mg Tablet
- Primidone (Mysoline®) 50 mg Tablets (Experimental): A single dose of Mysoline® 50 mg administered after an overnight fast of at least 10 hours.
  Interventions: Drug: Primidone (Mysoline®) 50 mg Tablet

INTERVENTIONS:
Drug: Primidone 50 mg Tablet — 50 mg tablet administered after an overnight fast of at least 10 hours.
  Arms: Primidone 50 mg Tablets
Drug: Primidone (Mysoline®) 50 mg Tablet — 50 mg tablet administered after an overnight fast of at least 10 hours.
  Other Names: Mysoline®
  Arms: Primidone (Mysoline®) 50 mg Tablets

SUMMARY:
The purpose of this study is to compare the bioequivalence of a test formulation of primidone tablets to an equivalent oral dose of the commercially available Mysoline®(primidone tablets) in adult subjects under fasting conditions.

DETAILED DESCRIPTION:
The purpose of this study is to compare the bioequivalence of a test formulation of primidone tablets to an equivalent oral dose of the commercially available Mysoline® (primidone tablets) in adult subjects under fasting conditions.

Twenty-two healthy, non-smoking, non-obese male and female volunteers at least 18 years of age will be randomly assigned in a crossover fashion to receive each of two primidone dosing regimens in sequence with a 14 day washout period between dosing periods. On the morning of Day 1, after an overnight fast of at least 10 hours, subjects will receive either a single oral dose of the test formulation, primidone (1 x 50 mg tablet) or a single oral dose of the reference formulation, Mysoline® (1 x 50 mg tablet). After a 14 day washout period, on the morning of Day 15 after an overnight fast, subjects will receive the alternate regimen. Blood samples will be drawn from all participants before dosing and for 72 hours post dose at times sufficient to adequately define the pharmacokinetics of primidone. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout the confinement portion of the study for adverse reactions to the study drugs and/or procedures. Blood pressure and heart rate will be obtained prior to dosing and at 3, 4, 6, 24 and 72 hours post-dose. All adverse events whether elicited by query, spontaneously reported or observed by clinic staff will be evaluated by the investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* at least 18 years of age
* weight must be 15% of ideal weight for height and frame
* subjects must be in good health and physical condition as determined by medical history
* subjects must read and sign consent form

Exclusion Criteria:

* history of treatment for alcoholism, substance abuse, or drug abuse within the last 24 months
* history of malignancy, stroke, diabetes, cardiac, renal or liver disease
* history of gastroesophageal reflux disease (GERD), malabsorption syndrome, colon cancer, chronic colitis, including Crohn's disease
* history of porphyria, hyperkinesia, respiratory diseases (eg. asthma, emphysema, difficulty breathing, pulmonary obstruction)
* females who pregnant or lactating
* history of hypersensitivity to primidone, barbiturates, and anticonvulsants
* sitting systolic blood pressure below 90mm Hg, or diastolic pressure below 50mm Hg (conditions upon screening which might contraindicate or require that caution be used in the administration of primidone)
* heart rate less than 50 beats per minute after a 5 minute rest
* treatment with any other investigational drug during the four weeks prior to initial dosing
* subjects who have donated blood within four weeks prior to the initial dosing
* subjects who smoke or use tobacco products or nicotine products. Three months abstinence is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-05; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Primidone 50 mg Tablets Then Mysoline® 50 mg Tablets: On the morning of Day 1 subjects received one tablet of the test formulation, primidone 50 mg, after an overnight fast of at least 10 hours, followed by a 14 day washout period. On the morning of Day 15 subjects received one tablet of the reference formulation, Mysoline® 50 mg, after an overnight fast of at least 10 hours.
- Mysoline® 50 mg Tablets Then Primidone 50 mg Tablets: On the morning of Day 1 subjects received one tablet of the reference formulation, Mysoline® 50 mg, after an overnight fast of at least 10 hours, followed by a 14 day washout period. On the morning of Day 15 subjects received one tablet of the test formulation, Primidone 50 mg, after an overnight fast of at least 10 hours.
Period: First Intervention
Arm/Group | Primidone 50 mg Tablets Then Mysoline® 50 mg Tablets | Mysoline® 50 mg Tablets Then Primidone 50 mg Tablets
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Washout Period of 14 Days
Arm/Group | Primidone 50 mg Tablets Then Mysoline® 50 mg Tablets | Mysoline® 50 mg Tablets Then Primidone 50 mg Tablets
Started | 11 | 11
Completed | 10 (adverse event- possible upper respiratory infection) | 11
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Second Intervention
Arm/Group | Primidone 50 mg Tablets Then Mysoline® 50 mg Tablets | Mysoline® 50 mg Tablets Then Primidone 50 mg Tablets
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Primidone 50 mg Tablets and Mysoline® 50 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 15, each subject received one tablet of either primidone 50 mg or Mysoline® 50 mg following an overnight fast of at least 10 hours.
Arm/Group | Primidone 50 mg Tablets and Mysoline® 50 mg Tablets
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 31.76 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 10
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma.
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to dose administration (0 hour) and at 0.33, 0.67, 1, 1.33, 1.67, 2, 2.33, 2.67, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 18, 24, 36, 48, 60 and 72 hours after drug administration.
Population: Plasma concentration data for 21 of 22 participants were used in the statistical analysis. One subject dropped from the study before Period II dosing due to an adverse event.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Primidone 50 mg Tablets: Each subject received one tablet of primidone 50 mg after an overnight fast of at least 10 hours.
- Mysoline® 50 mg Tablets: Each subject received one tablet of Mysoline® 50 mg after an overnight fast of at least 10 hours.
Arm/Group | Primidone 50 mg Tablets | Mysoline® 50 mg Tablets
Number analyzed (Participants) | 21 | 21
ng/mL | 1,165.92 (216.64) | 1,202.28 (273.28)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Primidone 50 mg Tablets | Mysoline® 50 mg Tablets
Number analyzed (Participants) | 21 | 21
ng-hr/mL | 27,893.57 (3,709.32) | 27,519.67 (3,606.54)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Primidone 50 mg Tablets | Mysoline® 50 mg Tablets
Number analyzed (Participants) | 21 | 21
ng-hr/mL | 31,162.82 (3,922.58) | 30,583.92 (3,786.58)

ADVERSE EVENTS:
Groups:
- Primidone 50 mg Tablets; Mysoline® 50 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 15, each subject received one tablet of either primidone 50 mg or Mysoline® 50 mg following an overnight fast.
Arm/Group | Primidone 50 mg Tablets | Mysoline® 50 mg Tablets
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 5/22 | 3/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primidone 50 mg Tablets (N=22) | Mysoline® 50 mg Tablets (N=21)
Confusion (Nervous system disorders) | 1 (1) | 1 (1)
Cramping (General disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 2 (2) | 0 (0)
Lightheadedness (Nervous system disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Near syncopal episode (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
Weakness (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days